CLINICAL TRIAL: NCT01317823
Title: Bishop Score and Transvaginal Ultrasound for Preinduction Cervical Assessment in Multiparas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BS_CL_02
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Failed Induction of Labor
Keywords: Multiparas, Bishop score, Cervical length, Cervical ripening

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bishop score (Active Comparator)
  Interventions: Other: Assessment of cervical status
- transvaginal ultrasound (Active Comparator)
  Interventions: Other: Assessment of cervical status

INTERVENTIONS:
Other: Assessment of cervical status — Assessment of cervical status based on Bishop score versus sonographically measured cervical length

SUMMARY:
To compare the ultrasonographic cervical length with the Bishop score in determining the administration of prostaglandin for preinduction cervical ripening in multiparous women at term.

ELIGIBILITY:
Inclusion Criteria:

* multiparous patients
* singleton pregnancy
* live fetus with vertex presentation
* intact amniotic membranes
* > 37 weeks gestation
* absence of labor
* no previous uterine surgical procedures

Exclusion Criteria:

* major congenital anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Successful labor induction | Eleven hours of initiating oxytocin on the fist day of induction
  Induction success was defined as an ability to achieve the active phase of labor corresponding to a cervical dilatation of ≥ 4 cm within 11 hours of initiating oxytocin (i.e., within 22 hours of the administration of a dinoprostone vaginal insert) on the first day of induction.

SECONDARY OUTCOMES:
the need for oxytocin induction, percentage of patients treated with prostagladins | After removing prostaglandin, the following day when an intravenous oxytocin infusion was started
  1. the interval from start of oxytocin to the active phase of labor
  2. the interval from start of oxytocin to delivery
  3. vaginal delivery within 24 hours of starting induction
  4. the incidence of cesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Hoon Park, MD, PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Obstetrics and Gynecology Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea